CLINICAL TRIAL: NCT01607762
Title: Comparison of Single-Dose Plasma and Blood Concentrations of Aripiprazole, Olanzapine, Quetiapine, Paliperidone and Risperidone After Capillary and Venous Blood Sample Collection
Brief Title: A Study to Compare Capillary and Venous Whole Blood and Plasma Concentrations of Five Antipsychotics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CR100831; INDIGO-APS-1001 (Other: Janssen Research & Development, LLC); 2011-006133-41 (EudraCT Number)
Record Dates: First submitted 2012-05-25; First posted 2012-05-30 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Healthy
Keywords: Healthy; Antipsychotics; Aripiprazole; Paliperidone; Risperidone; Quetiapine; Olanzapine
MeSH Terms: interventions — Aripiprazole; Quetiapine Fumarate; Olanzapine; Risperidone; Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort A: Aripiprazole (Experimental)
  Interventions: Drug: Aripiprazole
- Cohort B: Quetiapine (Experimental)
  Interventions: Drug: Quetiapine
- Cohort C: Olanzapine (Experimental)
  Interventions: Drug: Olanzapine
- Cohort D: Risperidone (Experimental)
  Interventions: Drug: Risperidone
- Cohort E: Paliperidone (Experimental)
  Interventions: Drug: Paliperidone

INTERVENTIONS:
Drug: Aripiprazole — Type= exact number, unit= mg, number= 5, form= tablet, route= oral administration. A single oral dose of a 5-mg aripiprazole tablet will be administered after an overnight fast.
  Arms: Cohort A: Aripiprazole
Drug: Quetiapine — Type= exact number, unit= mg, number= 100, form= tablet, route= oral administration. A single oral dose of two 50-mg quetiapine tablets will be administered after an overnight fast.
  Arms: Cohort B: Quetiapine
Drug: Olanzapine — Type= exact number, unit= mg, number= 5, form= tablet, route= oral administration. A single oral dose of a 5-mg olanzapine tablet will be administered after an overnight fast.
  Arms: Cohort C: Olanzapine
Drug: Risperidone — Type= exact number, unit= mg, number= 1, form= tablet, route= oral administration. A single oral dose of a 1-mg risperidone tablet will be administered after an overnight fast.
  Arms: Cohort D: Risperidone
Drug: Paliperidone — Type= exact number, unit= mg, number= 3, form= tablet, route= oral administration. A single oral dose of a 3-mg paliperidone tablet will be administered after an overnight fast.
  Arms: Cohort E: Paliperidone

SUMMARY:
The purpose of this study is to compare capillary (the smallest of a body's blood vessels) and venous whole blood and plasma concentrations of 5 antipsychotics after given of a single oral, immediate-release dose to healthy participants.

DETAILED DESCRIPTION:
This is a randomized (the study drug is assigned by chance), open-label (all people know the identity of the intervention), parallel-group (each group of patients will be treated at the same time), single-center study. Participants will be randomly assigned to 1 of 5 cohorts (groups) defined by the antipsychotic drug (aripiprazole, quetiapine, olanzapine, risperidone or paliperidone). Antipsychotics are drugs that are helpful in the treatment of psychosis and have a capacity to ameliorate thought disorders. Participants will enter the investigational site in the morning of Day -1 and stay until the morning of Day 2. Participants will return to the study site for subsequent assessments as per study's schedule. The total study length for a participant is approximately 26 days, except for participants receiving aripiprazole for whom the total study length is approximately 39 days.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (weight [kg]/height2 [m]2) between 17 and 35 kg/m2 (inclusive), and body weight not less than 50 kg
* If a woman, must be postmenopausal, surgically sterile, abstinent, or, if sexually active, be practicing an effective method of birth control before entry and throughout the study
* If a woman, must have negative pregnancy test at screening
* If a man, must agree to use an adequate contraception method as deemed appropriate by the investigator and to not donate sperm during the study and for 3 months after receiving the study drug
* Blood pressure between 90 and 140 mmHg systolic, inclusive, and no higher than 90 mmHg diastolic

Exclusion Criteria:

* History of or current clinically significant medical illness or condition that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Clinically significant abnormal values for laboratorial tests
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements), except for paracetamol (acetaminophen), oral contraceptives and hormonal replacement therapy, within 14 days before the study drug administration is scheduled
* Positive test for alcohol or drugs of abuse at screening
* Unable to swallow solid, oral dosage forms whole with the aid of water (participants may not chew, divide, dissolve, or crush the study drug)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2012-02; Primary Completion 2012-04 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Aripiprazole concentration in venous and capillary plasma, venous and capillary whole blood | 16 time points over 408 hours postdose
Quetiapine concentration in venous and capillary plasma, venous and capillary whole blood | 12 time points over 108 hours postdose
Olanzapine concentration in venous and capillary plasma, venous and capillary whole blood | 12 time points over 108 hours postdose
Risperidone concentration in venous and capillary plasma, venous and capillary whole blood | 12 time points over 108 hours postdose
Paliperidone concentration in venous and capillary plasma, venous and capillary whole blood | 12 time points over 108 hours postdose
Dehydroaripiprazole concentration in venous and capillary plasma, venous and capillary whole blood | 16 time points over 408 hours postdose
9 hydroxy-risperidone concentration in venous and capillary plasma, venous and capillary whole blood | 12 time points over 108 hours postdose

SECONDARY OUTCOMES:
Incidence of adverse events as a measure of safety and tolerability | Approximately 26 days (Cohorts B, C, D, E), and approximately 39 days (Cohort A)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Merksem, Belgium